CLINICAL TRIAL: NCT00566514
Title: The Role of D-RIbose in Patients Diagnosed With Fibromyalgia
Brief Title: The Role of Ribose in Patients Diagnosed With Fibromyalgia
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol Under Review
Sponsor: Bioenergy Life Science, Inc. (Industry)
Responsible Party: Jacob Teitelbaum, MD, The Annapolis Center for Effective CFS/Fibromyalgia Therapies
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 200604-7
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; ribose; d-ribose; dextrose
MeSH Terms: conditions — Fibromyalgia | interventions — Ribose; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): D-ribose 5 grams TID orally
  Interventions: Dietary Supplement: D-ribose
- 2 (Placebo Comparator): Dextrose 5 grams TID
  Interventions: Other: dextrose

INTERVENTIONS:
Dietary Supplement: D-ribose — 5 grams administered orally TID
  Other Names: Corvalen
  Arms: 1
Other: dextrose — 5 grams orally TID
  Arms: 2

SUMMARY:
The purose of this research study is to determine the potential benefit of D-ribose, a nutritional supplement (a sugar), versus a placebo (another sugar) in people with fibromyalgia.

DETAILED DESCRIPTION:
Two hundred to three hundred subjects (equally distribued between placebo and D-ribose) between 18-78 years of age will comprise this study. The final numbers enrolled will depend upon obtaining approximately 100 subjects that can display a high degree of compliance to TID dosing with approximately equal balance between the active and placebo arms.

ELIGIBILITY:
Inclusion Criteria:

* previous diagnosis of fibromomyalgia by a MD
* Has been diagnosed with fibromyalgia and are over 18 years of age
* Does live in the United States

Exclusion Criteria:

* does NOT have severe medication/chemical/supplement sensitivities
* does NOT have insulin dependent diabetes or other severe illnesses (cancer, hepatitis, congestive heart failure)
* does NOT have rheumatoid arthritis or gout
* previous use of ribose

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-07 (Estimated); Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Significant reduction in symptoms of pain and fatigue | 3 weeks

SECONDARY OUTCOMES:
Demonstrate an improvement in ones quality of life | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Teitelbaum, MD, Principal Investigator — The Annapolis Center for Effective CFS/Fibromyalgia Therapies; Kent Holtorf, MD, Principal Investigator — Hormone and Longevity Medical Center
Locations (1):
- Bioenergy Life Science, Inc., Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Teitelbaum JE, Johnson C, St Cyr J. The use of D-ribose in chronic fatigue syndrome and fibromyalgia: a pilot study. J Altern Complement Med. 2006 Nov;12(9):857-62. doi: 10.1089/acm.2006.12.857. PMID 17109576